CLINICAL TRIAL: NCT06302803
Title: Effects of Modified Intermittent Eating Strategy on Weight Loss and Cardiometabolic Risk Factors in Obese Adults: a Randomized Clinical Trial
Brief Title: Modified Intermittent Eating on Weight Loss (INTEREST-3 Trial)
Acronym: INTEREST-3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NFEC-2024-033
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Obesity
Keywords: Obesity; Time restricted eating; Intermittent Fasting; Modified Intermittent Eating strategy; Calorie restriction; Weight loss
MeSH Terms: conditions — Obesity; Intermittent Fasting; Weight Loss | interventions — Caloric Restriction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The mTRE group (Experimental): Participants in the mTRE group will be instructed to eat during a window of 8 h (8 am to 4 pm) 5 days and fast (approximately 500-600 kcal per day) 2 days per week.
  Interventions: Behavioral: Intermittent fasting plus time-restricted eating
- The CR group (Experimental): Participants will follow receive a diet of 1500-1800kcal/d for men and 1200-1500kcal/d for women, without restriction on eating time.
  Interventions: Behavioral: Calorie restriction
- Control (No Intervention): usual health care

INTERVENTIONS:
Behavioral: Intermittent fasting plus time-restricted eating — Participants in the mTRE group will be instructed to eat during a window of 8 h (8 am to 4 pm) 5 days and fast (approximately 500-600 kcal per day) 2 days per week.
  Other Names: mTRE
  Arms: The mTRE group
Behavioral: Calorie restriction — Participants will follow receive a diet of 1500-1800kcal/d for men and 1200-1500kcal/d for women, without restriction on eating time.
  Other Names: CR
  Arms: The CR group

SUMMARY:
Calorie restriction (CR) is the most important treatment for weighting loss. In recent years, two novel types of intermittent fasting recently have gained more attention: the 5:2 diet and time-restricted eating (TRE). TRE requires individuals to eat in a specified number of hours per day (typically 4 to 10 hours) without energy intake restriction. The 5:2 diet involves 5 feast days and 2 fast days per week; participants eat ad libitum without restriction on feast days while 25% of energy needs (approximately 500-800 kcal per day) are consumed on fast days. However, the effects of dietary strategy of intermittent fasting plus time-restricted eating (modified time-restricted eating: TRE 5 days and fasting 2days per week) on weight loss and cardiometabolic risk factors in obese adults have not been proved. This randomized controlled trial aimed to evaluate the effect of modified time-restricted eating (mTRE) and CR on weight loss and cardiometabolic risk factors in obese adults compared to usual health care over 12 months.

DETAILED DESCRIPTION:
Obesity is becoming a major global public health issue. Calorie restriction (CR) is the most important treatment for weighting loss. In recent years, two novel types of intermittent fasting recently have gained more attention: the 5:2 diet and time-restricted eating (TRE). TRE requires individuals to eat in a specified number of hours per day (typically 4 to 10 hours) without energy intake restriction. The 5:2 diet involves 5 feast days and 2 fast days per week; participants eat ad libitum without restriction on feast days while 25% of energy needs (approximately 500-800 kcal per day) are consumed on fast days. However, the effects of dietary strategy of intermittent fasting plus time-restricted eating (modified time-restricted eating: TRE 5 days and fasting 2days per week) on weight loss and cardiometabolic risk factors in obese adults have not been proved. This randomized controlled trial aimed to evaluate the effect of modified time-restricted eating (mTRE) and CR on weight loss and cardiometabolic risk factors in obese adults compared to usual health care over 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Man or women aged 18-75 years;
2. Body mass index (BMI)of 28.0 to 45.0 kg/m2;

Exclusion Criteria:

1. History of HIV, hepatitis B or C (self-report) or active pulmonary tuberculosis;
2. Diagnosis of type 1 and type 2 diabetes;
3. History of malignant tumors;
4. Serious liver dysfunction or chronic kidney disease (AST or ALT > 3 times the upper limit of normal, or eGFR<30 ml/min/1.73 m2);
5. History of serious cardiovascular or cerebrovascular disease (angina, myocardial infarction or stroke) in the past 6 months;
6. History of severe gastrointestinal diseases or gastrointestinal surgery in the past 12 months;
7. History of Cushing's syndrome, hypothyroidism, acromegaly, hypothalamic obesity;
8. Being a smoker or having been a smoker in the 3 months prior to their screening visit;
9. Taking medications affecting weight or energy intake/energy expenditure in the last 6 months, including weight loss medications, antipsychotic drugs or other medications as determined by the study physician;
10. Currently participating in weight loss programs or weight change in the past 3 months (> 5% current body weight) ;
11. Women who are pregnant or plan to become pregnant;
12. Patients who cannot be followed for 24 months (due to a health situation or migration);
13. Patients who are unwilling or unable to give informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2024-04-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in body weight over 12 months | Baseline to months 12
  Change in body weight over 12 months

SECONDARY OUTCOMES:
Change in body mass index （BMI） | Baseline to months 12
  body mass index : the weight in kilograms divided by the square of the height in meters.The higher scores mean a worse outcome.
Change in waist circumference | Baseline to months 12
  Wrap a tape measure around the waist at the level of the navel.
Change in body fat composition meassured by DEXA | Baseline to months 12
  Body composition is meassured by dual-energy X-ray absorptiometry scans
Change in liver fat | Baseline to months 12
  Liver fat is assessed by liver Fibroscan
Change in systolic blood pressure | Baseline to months 12
  blood pressure
Change in diastolic blood pressure | Baseline to months 12
  blood pressure
Change in concentration of serum triglyceride | Baseline to months 12
  the contents of serum triglyceride
Change in concentration of serum total cholesterol | Baseline to months 12
  the contents of serum total cholesterol
Change in concentration of serum LDL-c | Baseline to months 12
  the contents of Low Density Lipoprotein
Change in concentration of HbA1c | Baseline to months 12
  the contents of Glycated hemoglobin
Change in insulin sensitivity | Baseline to months 12
  Insulin sensitivity is assessed by HOMA-IR (Homeostatic Model Assessment for Insulin Resistance).
Change in β cell function | Baseline to months 12
  β cell function is assessed by HOMA-B
Change in arterial stiffness measured by pulse wave velocity | Baseline to months 12
  arterial stiffness is measured by pulse wave velocity (PWV)
Change in depression score measured by the Patient Health Questionnaire-9 | Baseline to months 12
  Depression is measured by the Patient Health Questionnaire-9 (PHQ-9). The maximum value is 27, and the minimum value is 0 . The higher scores mean a worse outcome.
Change in quality of sleep score measured by the Pittsburgh sleep quality index | Baseline to months 12
  Quality of sleep is measured by the Pittsburgh sleep quality index (PSQI). The maximum value is 21, and the minimum value is 0 . The higher scores mean a worse outcome.
Change in quality of life score measured by the 12-item Short-Form Health Survey Questionnaire | Baseline to months 12
  Quality of life is measured by the 12-item Short-Form Health Survey Questionnaire (SF-12). The maximum value is 100, and the minimum value is 0 . The higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Huijie Zhang, MD. PhD., Principal Investigator — Department of Endocrinology and Metabolism, Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No